CLINICAL TRIAL: NCT06290128
Title: A Phase 3, Double-blind, Placebo-controlled Study Evaluating Efficacy and Safety of Riliprubart in Participants With Refractory Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: A Study to Test the Effects and Safety of Riliprubart in People With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) for Which the Usual Treatments do Not Work
Acronym: MOBILIZE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17236; U1111-1295-5755 (Registry Identifier: ICTRP); 2023-506503-26 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Polyneuropathy, Inflammatory Demyelinating, Chronic
Keywords: Autoimmune Diseases, Neurologic; Autoimmune Disorders, Nervous System; Peripheral Nerves Disease; Nervous System Diseases; Neurologic Disorders; Neurological Disorders; Complement Inhibitor; Complement Inhibitors
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Autoimmune Diseases of the Nervous System; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This is a double-blind treatment in part A and open-label treatment in Part B.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riliprubart Arm (Experimental): Riliprubart for 24 weeks followed by open-label extension phase with riliprubart for 24 weeks
  Interventions: Drug: Riliprubart; Drug: Placebo
- Placebo Arm (Placebo Comparator): Placebo for 24 weeks followed by open-label extension phase with riliprubart for 24 weeks
  Interventions: Drug: Riliprubart; Drug: Placebo

INTERVENTIONS:
Drug: Riliprubart — Pharmaceutical form: Solution Route of administration: IV Infusion
  Other Names: SAR445088
Drug: Placebo — Pharmaceutical form: Solution Route of administration: IV Infusion
Drug: Riliprubart — Pharmaceutical form: Solution Route of administration: SC Injection
  Other Names: SAR445088
Drug: Placebo — Pharmaceutical form: Solution Route of administration: SC Injection

SUMMARY:
The purpose of the study is to evaluate efficacy of riliprubart compared to placebo in adult participants with CIDP whose disease is refractory to standard of care. The study duration will be for a maximum of 111 weeks including screening, treatment phases, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

-Participant must have CIDP or possible CIDP criteria, based on European Academy of Neurology (EAN)/ Peripheral Nerve Society (PNS) Task Force CIDP guidelines, second revision (2021).

* Participant must have either typical CIDP, or one of the following two CIDP variants: motor CIDP (including motor predominant), multifocal CIDP (also known as Lewis Sumner Syndrome). Diagnosis must be confirmed by the adjudication committee.
* Participant must be refractory to either immunoglobulin therapy or corticosteroid therapy, as defined below.

  * Immunoglobulinrefractory subgroup: Historic evidence of failure or inadequate response to immunoglobulin therapy prior to screening, defined as no clinically meaningful improvement or persistent INCAT score ≥2 after a minimum of:

    * One dose of IVIg of 2 g/kg, followed by a second dose of 2 g/kg or two doses of 1 g/kg, with a separation of approximately 3 weeks between doses (each dose can be divided over 2 to 5 days), as indicated in the EAN/PNS 2021 guidelines OR
    * SCIg maintenance therapy with at least 0.2 g/kg weekly for 5 weeks
  * Corticosteroidrefractory subgroup:

Historic evidence of failure or inadequate response to corticosteroid therapy prior to screening, defined as no clinically meaningful improvement or persistent INCAT score ≥2 after a minimum of 12 weeks of corticosteroid therapy. Corticosteroid regimen can be daily oral prednisone/prednisolone, at least 60 mg, equivalent to methylprednisolone 48 mg, tapered over 6 to 8 months, or alternative regimens, e.g. pulsed high-dose corticosteroid treatment (40 mg/day oral dexamethasone or 500 mg/day IV methylprednisolone, each daily for 4 days per month for 6 months), as indicated in the EAN/PNS 2021 guidelines A clinically meaningful improvement is defined as one or more of the following:

* A ≥1 point decrease in adjusted INCAT disability score
* An increase in IRODS centile score ≥4 points
* An increase in MRC Sum score ≥3 points
* An improvement in hand grip strength of ≥8 kilopascals or
* Equivalent improvement based on information from medical records and per the Investigator's judgment

  * Participant has an adjusted INCAT score of 2 to 9

    --(a score of 2 should be exclusively from the leg disability component of INCAT).
  * Any allowed immunosuppressant drugs (azathioprine, cyclosporine, or mycophenolate mofetil) have been taken for ≥6 months at a stable dose for ≥3 months prior to Screening
  * Participant may be receiving low-dose oral corticosteroids (≤20 mg/day of prednisone [or equivalent dose for other oral corticosteroids]), but only if taken at a stable dose for ≥3 months prior to Screening
  * Participant must have active disease, defined by a CIDP disease activity score (CDAS) of ≥ 2 points at Screening
  * Participant must have documented vaccinations against encapsulated bacterial pathogens given within 5 years prior to Day 1 or initiated a minimum of 14 days prior to first dose of study intervention
  * All participants must agree to use contraception methods during and after the study as required.
  * Contraceptive use by men and women participating in the study should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    * Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 55 weeks after the last dose of study medication:
* Refrain from donating or cryopreserving sperm PLUS
* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception/barrier as detailed below:

  ---- A male condom and an additional highly effective contraceptive method as described in the protocol.

  -- A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:
* Is a woman of nonchildbearing potential (WONCBP) as defined by the protocol OR
* Is a woman of childbearing potential (WOCBP) and agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), as described in Appendix 10.4 Contraception and barrier guidance during the study intervention period (to be effective before starting the intervention) and for at least 55 weeks after the last administration of study intervention and agrees not to donate or cryopreserve eggs (ova, oocytes) for the purpose of reproduction during this period.

  * Body weight at Screening of 35 kg to 154 kg (77 to 340 lbs), inclusive

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Polyneuropathy of other causes, including but not limited to: hereditary demyelinating neuropathies, neuropathies secondary to infection or systemic disease, diabetic neuropathy, drug- or toxin-induced neuropathies, multifocal motor neuropathy, polyneuropathy related to Immunoglobulin M (IgM) monoclonal gammopathy, POEMS syndrome, and lumbosacral radiculoplexus neuropathy.
* Sensory CIDP, Distal CIDP and focal CIDP variants.
* Any other neurological or systemic disease that can cause symptoms and signs interfering with treatment or outcome assessments
* Poorly controlled diabetes (HbA1c >7%)
* Serious infections requiring hospitalization within 30 days prior to Screening and any active infection requiring treatment during screening or presence of a condition that may predispose the participant to increased risk of infection (eg, medical history such as known immunodeficiency or history of recurrent infections)
* Clinical diagnosis of Systemic Lupus Erythematosus (SLE) or family history of SLE. For a participant with an antinuclear antibody (ANA) titer ≥1:160 and a positive anti-double-stranded DNA (anti-dsDNA) at Screening, SLE diagnosis must be ruled out prior to enrollment.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study. Specifically, history of any hypersensitivity reaction to riliprubart or its components or of a severe allergic or anaphylactic reaction to any humanized or murine monoclonal antibody.
* Any other clinically meaningful medical history or ongoing medical condition (as determined by the Investigator at Screening) that might impact benefitrisk assessment, jeopardize the safety of the participant, or compromise the quality of the data collected in this study; or history or presence of other significant concomitant illness that would adversely affect participation in this study, per Investigator's judgment.
* Documented history of attempted suicide over the 6 months prior to the Screening visit, presence of suicidal ideation of category 4 or 5 on CSSRS during screening, OR if in the Investigator's judgment, the participant is at risk for a suicide attempt.
* Evidence of CIDP worsening within the 6 weeks following a prior vaccination that, in the opinion of the Investigator, constituted a relapse
* Recent or planned major surgery that could confound the results of the trial or put the participant at undue risk
* Participant has received immunoglobulins (IVIg or SCIg) within 8 weeks prior to Screening
* Treatment with plasma exchange within the 8 weeks prior to Screening
* Prior treatment with riliprubart
* Prior treatment with (any time) with highly immunosuppressive/chemotherapeutic medications with sustained effects, eg, mitoxantrone, alemtuzumab, cladribine
* Prior treatment (any time) with total lymphoid irradiation or bone marrow transplantation
* Prior treatment with B-cell-depleting agents such as rituximab within 6 months prior to riliprubart dosing, or until return of B-cells counts to normal levels, whichever is longer
* Use of any specific complement system inhibitor (eg, eculizumab) within 12 weeks or 5 times the halflife of the product, whichever is longer, prior to Screening
* Treatment within 6 months prior to dosing with immunosuppressive/ chemotherapeutic medications, such as cyclophosphamide, methotrexate, tacrolimus, interferon, or tumor necrosis factor (TNF)α inhibitors. Certain immunosuppressants commonly used in CIDP (azathioprine, cyclosporine, or mycophenolate mofetil) are allowed, as indicated under inclusion criterion.
* Any vaccination received within 28 days prior to dosing (with few exceptions to be confirmed at screening)
* Participation in another clinical trial with an investigational drug or receipt of an investigational product within 12 weeks or 5 times the halflife of the product, whichever is longer, prior to Screening
* Any screening laboratory values outside normal limits or abnormal ECG considered in the Investigator's judgment to be clinically significant in the context of this trial.
* Positive result of any of the following tests:

  * hepatitis B surface antigen (HBsAg)
  * antihepatitis B core antibodies (anti-HBc Ab) (unless anti-hepatitis B surface antibodies [antiHBs Ab] are also positive, indicating natural immunity)
  * antihepatitis C virus (antiHCV) antibodies
  * antihuman immunodeficiency virus 1 and 2 (antiHIV1 and antiHIV2) antibodies
* Pregnancy, defined as a positive result of a highly sensitive urine or serum pregnancy test, or lactation
* Accommodation in an institution because of regulatory or legal order; eg, imprisoned or legally institutionalized
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or potential risk for noncompliance to study procedures
* Participants are employees at the clinical study site or other individuals directly involved in the conduct of the study, or immediate family member of such individuals
* Any country related specific regulation that would prevent the participant from entering the study
* Treatment with efgartigimod within 8 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing a response | Baseline to week 24
  A response is defined as a decrease of ≥1 point from baseline in adjusted INCAT disability score at Week 24.
Percentage of participants randomized to riliprubart with lasting response | Baseline to week 48
  Lasting response is defined as a decrease of ≥1 point in adjusted INCAT disability score at week 48 versus baseline.
Percentage of participants randomized to placebo who experience a response | Week 24 to week 48
  A response is defined as a decrease of ≥1 point in adjusted INCAT disability score at Week 48 versus week 24.

SECONDARY OUTCOMES:
Change from baseline in Inflammatory Raschbuilt Overall Disability Scale (IRODS) score | Baseline to week 24
Change from baseline in adjusted inflammatory neuropathy cause and treatment (INCAT) disability score | Baseline to week 24
Change from baseline in grip strength (kilopascals; dominant hand) | Baseline to week 24
Change from baseline in Medical Research Council Sum Score (MRC-SS) | Baseline to week 24
Percentage of participants refractory to immunoglobulins experiencing a response | Baseline to week 24
  A response is defined as a decrease of ≥1 point from baseline in adjusted INCAT disability score at Week 24
Change from baseline in the EuroQol 5 Dimension, 5-Level Health Scale (EQ-5D-5L) | Baseline to week 24
Change from baseline in the Rasch-built modified fatigue severity scale (RT-FSS) | Baseline to week 24
Number of participants with treatment emergent adverse events (TEAEs), including serious adverse events (SAEs) and adverse events of special interest (AESIs) for Part A | Baseline to week 24
Incidence and titer of anti-riliprubart antibodies (ADA) | Baseline to week 24
Number of participants with TEAEs, including Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) for Part B | Week 24 to week 111
Incidence and titer of anti-riliprubart antibodies | Week 24 to week 111
Change from baseline in I RODS score | Baseline to week 48
Change from baseline in adjusted INCAT score | Baseline to week 48
Change from baseline in grip strength (kilopascals; dominant hand) | Baseline to week 48
Change from baseline in MRC-SS | Baseline to week 48
Change from baseline in EQ-5D-5L score | Baseline to week 48
Change from baseline in RT-FSS | Baseline to week 48
Percentage of participants randomized to riliprubart who experience a response at Week 48 without prior response in Part A (delayed response) | Baseline to week 48
  A delayed response is defined as a decrease of ≥1 point in adjusted INCAT disability score at Week 48 versus baseline.

CONTACTS AND LOCATIONS:
Locations (116):
- United States (20):
  - Alabama Neurology Associates- Site Number : 8400019, Homewood, Alabama
  - USC Norris Comprehensive Cancer Center- Site Number : 8400002, Los Angeles, California
  - University of California Irvine - Manchester Pavilion- Site Number : 8400007, Orange, California
  - Yale University School of Medicine- Site Number : 8400018, New Haven, Connecticut
  - NorthShore University Health System - Glenbrook Hospital- Site Number : 8400024, Glenview, Illinois
  - University of Kansas Medical Center- Site Number : 8400010, Kansas City, Kansas
  - NeuroMedical Clinic of Central Louisiana- Site Number : 8400031, Alexandria, Louisiana
  - Ochsner Medical Center - Jefferson Highway- Site Number : 8400030, New Orleans, Louisiana
  - Johns Hopkins Hospital- Site Number : 8400015, Baltimore, Maryland
  - Henry Ford Hospital- Site Number : 8400025, Detroit, Michigan
  - Michigan State University- Site Number : 8400038, East Lansing, Michigan
  - Washington University School of Medicine - Siteman Cancer Center- Site Number : 8400037, St Louis, Missouri
  - Hospital for Special Surgery- Site Number : 8400041, New York, New York
  - Columbia University Irving Medical Center- Site Number : 8400003, New York, New York
  - University of Cincinnati Medical Center- Site Number : 8400020, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 8400033, Cleveland, Ohio
  - Penn Medicine: University of Pennsylvania Health System- Site Number : 8400022, Philadelphia, Pennsylvania
  - Austin Neuromuscular Center- Site Number : 8400040, Austin, Texas
  - University of Vermont Medical Center- Site Number : 8400012, Burlington, Vermont
  - University of Virginia- Site Number : 8400023, Charlottesville, Virginia
- Argentina (3):
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
- Investigational Site Number : 0560001, Leuven, Belgium
- Brazil (5):
  - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo- Site Number : 0760012, Vitória, Espírito Santo
  - Hospital Sao Rafael- Site Number : 0760011, Salvador, Estado de Bahia
  - Hospital Moinhos de Vento- Site Number : 0760003, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto- Site Number : 0760007, Ribeirão Preto, São Paulo
  - PSEG Centro de Pesquisa Clínica- Site Number : 0760009, São Paulo
- Bulgaria (2):
  - Investigational Site Number : 1000002, Blagoevgrad
  - Investigational Site Number : 1000001, Pleven
- Investigational Site Number : 1240001, Québec, Quebec, Canada
- Chile (3):
  - Investigational Site Number : 1520003, Lo Barnechea, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- China (16):
  - Investigational Site Number : 1560013, Beijing
  - Investigational Site Number : 1560010, Beijing
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560016, Beijing
  - Investigational Site Number : 1560009, Changsha
  - Investigational Site Number : 1560011, Chengdu
  - Investigational Site Number : 1560002, Fuzhou
  - Investigational Site Number : 1560012, Guangzhou
  - Investigational Site Number : 1560007, Guangzhou
  - Investigational Site Number : 1560014, Hangzhou
  - Investigational Site Number : 1560008, Jinan
  - Investigational Site Number : 1560015, Nanchang
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560003, Wuhan
  - Investigational Site Number : 1560006, Wuhan
  - Investigational Site Number : 1560004, Xi'an
- Czechia (3):
  - Investigational Site Number : 2030004, Brno
  - Investigational Site Number : 2030003, Hradec Králové
  - Investigational Site Number : 2030002, Pardubice
- Denmark (2):
  - Investigational Site Number : 2080002, Aarhus
  - Investigational Site Number : 2080001, Copenhagen
- France (4):
  - Investigational Site Number : 2500001, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500003, Lille
  - Investigational Site Number : 2500002, Marseille
  - Investigational Site Number : 2500004, Paris
- Germany (4):
  - Massachusetts General Hospital- Site Number : 8400009, Berlin, Massachusetts
  - Investigational Site Number : 2760001, Bad Homburg
  - Investigational Site Number : 2760003, Giessen
  - Investigational Site Number : 2760006, Tübingen
- Greece (3):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000003, Larissa
  - Investigational Site Number : 3000001, Thessaloniki
- Italy (9):
  - Investigational Site Number : 3800001, Milan, Milano
  - Investigational Site Number : 3800009, Rozzano, Milano
  - Investigational Site Number : 3800006, Rome, Roma
  - Investigational Site Number : 3800002, Rome, Roma
  - Investigational Site Number : 3800008, Rome, Roma
  - Investigational Site Number : 3800007, Messina
  - Investigational Site Number : 3800003, Palermo
  - Investigational Site Number : 3800005, Pavia
  - Investigational Site Number : 3800004, Pisa
- Japan (10):
  - Investigational Site Number : 3920006, Sayama, Osaka
  - Investigational Site Number : 3920005, Kawagoe, Saitama
  - Investigational Site Number : 3920014, Yaizu, Shizuoka
  - Investigational Site Number : 3920011, Bunkyo, Tokyo
  - Investigational Site Number : 3920008, Kodaira, Tokyo
  - Investigational Site Number : 3920001, Chiba
  - Investigational Site Number : 3920003, Fukuoka
  - Investigational Site Number : 3920009, Saga
  - Investigational Site Number : 3920013, Tokyo
  - Investigational Site Number : 2500005, Toyama
- Mexico (3):
  - Investigational Site Number : 4840003, Guadalajara, Jalisco
  - Investigational Site Number : 4840005, Culiacán, Sinaloa
  - Investigational Site Number : 4840002, Veracruz
- Netherlands (2):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280002, Rotterdam
- Poland (3):
  - Investigational Site Number : 6160006, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160002, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6160003, Rzeszów, Podkarpackie Voivodeship
- Portugal (4):
  - Investigational Site Number : 6200005, Coimbra
  - Investigational Site Number : 6200004, Lisbon
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200003, Matosinhos Municipality
- South Korea (3):
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (7):
  - Investigational Site Number : 7240008, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240007, Bilbao, Basque Country
  - Investigational Site Number : 7240001, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240006, Majadahonda, Madrid
  - Investigational Site Number : 7240003, Pamplona, Navarre
  - Investigational Site Number : 7240005, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240002, Valencia
- Investigational Site Number : 7520001, Stockholm, Sweden
- Taiwan (3):
  - Investigational Site Number : 1580003, Kaohsiung City
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580002, Taipei
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920002, Bursa
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920004, Istanbul
  - Investigational Site Number : 7920003, Konya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18156 (Vitalize) & EFC17236 (MOBILIZE) CIDP website-for potential participants — https://www.sanofistudies.com/G4SB
- See also: EFC17236 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25645&tenant=MT_SNY_9011